CLINICAL TRIAL: NCT05738928
Title: Microbiological Profile of Ventilator Associated Pneumonia in Respiratory Intensive Care Unit of Assiut University Hospital
Brief Title: Microbiological Profile of VAP Patients in Respiratory ICU
Acronym: VAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Abdelhameed Hassan Ali, Doctor, Assiut University
Other Study IDs: Microbiological profile of VAP
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: VAP - Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood and sputum culture — Noninvasive sampling ( Endo Tracheal Aspiration) for staining and culture. Blood culture .

SUMMARY:
Identification of the microbial profile of Ventilator associated pneumonia causing microorganisms among Respiratory ICU patients .

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is one of the common serious infectious diseases encountered in the intensive care unit (ICU), which highly affects the healthcare cost and patient prognosis.

All-cause of mortality associated with VAP has been reported to range from 20% to 50%.

The etiology of VAP and their antimicrobial susceptibility pattern varies with different patient populations and types of ICUs.

VAP may be caused by a wide spectrum of bacterial pathogens, which may be polymicrobial and are rarely due to viral or fungal pathogens in immune-competent hosts.

Common etiologic agents are Gram-negative bacilli such as Pseudomonas aeruginosa, Escherichia coli, Klebsiella pneumoniae, and Acinetobacter spp. and Staphylococcus aureus among Gram-positive cocci.

Due to the increased incidence of MDR organisms in Intensive Care Units (ICUs), early and correct diagnosis of VAP is mandatory for optimal antibiotic therapy. The frequency of specific MDR pathogens causing VAP varies in hospitals, patient populations. Also varies according underlying disease.

this study will be conducted in respiratory intensive care unit, chest disease and tuberculosis department at Assiut university hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanically ventilated patient who developed pneumonia after48 hours after endotracheal intubation.
2. Age > 18 years.

Exclusion Criteria:

1. Patients with clinical and radiological signs suggestive of pneumonia before intubation (community acquired pneumonia or hospital acquired pneumonia)
2. Patients age ≤18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age more than 18 years.
  Mechanically ventilated patient who developed pneumonia after48 hours after endotracheal intubation.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Microbiological profile of ventilator associated pneumonia in Respiratory ICU in Assiut University Hospital. | 1 year
  Identify the microbial profile of VAP causing microorganisms among ICU patients, antimicrobial susceptibility patterns among the frequently isolated organisms and resistant strains.

CONTACTS AND LOCATIONS:
Overall Officials: mohammed M Abdelhadi, PhD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided